CLINICAL TRIAL: NCT05625477
Title: A Multicenter, Randomized, Double-Blind, Parallel-Controlled, Dose-Finding Phase II Study to Compare the Anti-tetanus Neutralizing Antibody Titers and Safety of TNM002 Injection With Human Tetanus Immunoglobulin or Placebo Following a Single Intramuscular Injection in Chinese Adult Volunteers
Brief Title: Study to Compare the Anti-tetanus Neutralizing Antibody Titers and Safety of TNM002 Injection With Human Tetanus Immunoglobulin or Placebo in Adult Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhuhai Trinomab Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TNM002-P2-CH01
Record Dates: First submitted 2022-11-11; First posted 2022-11-23 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2023-05

CONDITIONS: Tetanus
MeSH Terms: conditions — Tetanus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- TNM002 low dose (Experimental): Participants receive a single intramuscular injection of TNM002 with low dose on Day 1
  Interventions: Biological: TNM002 (low dose)
- TNM002 medium dose (Experimental): Participants receive a single intramuscular injection of TNM002 with medium dose on Day 1
  Interventions: Biological: TNM002 (medium dose)
- TNM002 high dose (Experimental): Participants receive a single intramuscular injection of TNM002 with high dose on Day 1
  Interventions: Biological: TNM002 (high dose)
- Human Tetanus Immunoglobulin (HTIG) (Active Comparator): Participants receive a single intramuscular injection of human tetanus immunoglobulin 250 IU on Day 1
  Interventions: Biological: HTIG
- Placebo (Placebo Comparator): Participants receive a single intramuscular injection of placebo on Day 1
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TNM002 (low dose) — Single dose of TNM002 administered by intramuscular injection
  Arms: TNM002 low dose
Biological: TNM002 (medium dose) — Single dose of TNM002 administered by intramuscular injection
  Arms: TNM002 medium dose
Biological: TNM002 (high dose) — Single dose of TNM002 administered by intramuscular injection
  Arms: TNM002 high dose
Biological: HTIG — Single dose of HTIG administered by intramuscular injection
  Arms: Human Tetanus Immunoglobulin (HTIG)
Biological: Placebo — Single dose of placebo administered by intramuscular injection
  Arms: Placebo

SUMMARY:
The primary objective is to compare the anti-tetanus neutralizing antibody titers of TNM002 Injection with human tetanus immunoglobulin (HTIG) following a single intramuscular (IM) injection in Chinese adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese male or female adults aged ≥ 18 years;
2. Healthy volunteers or volunteers with stable chronic diseases;
3. Volunteers who provide signed written informed consent form.

Exclusion Criteria:

1. History of allergy to the investigational product, human immunoglobulin preparation or any component of other therapeutic monoclonal immunoglobulins;
2. Any clinically significant chronic or acute medical condition that makes the volunteer unsuitable for participation;
3. History of alcohol or other substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2022-05-29 (Actual); Study Completion 2022-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jie Hou, Principal Investigator — Peking University Care Luzhong Hospital
Locations (4):
- China (4):
  - The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - PKUCare Luzhong Hospital, Zibo, Shandong
  - Yunnan Provincial Hospital of Traditional Chinese Medicine, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 240 adult participants were recruited from 4 study sites in China, from 18 April 2022 to 27 May 2022.
Pre-assignment Details: There were 402 participants excluded from the trial before assignment to any arm, primarily due to failure to meet eligibility criteria (369 participants) and other (33).
Groups:
- TNM002 5 mg; TNM002 10 mg; TNM002 15 mg; Placebo: Double blind, a single intramuscular injection on Day 1
- HTIG: Double blind, a single intramuscular injection of Human Tetanus Immunoglobulin (HTIG) 250 IU on Day 1
Period: Overall Study
Arm/Group | TNM002 5 mg | TNM002 10 mg | TNM002 15 mg | HTIG | Placebo
Started | 61 | 61 | 29 | 59 | 30
Completed | 58 | 59 | 28 | 58 | 30
Not Completed | 3 | 2 | 1 | 1 | 0
Not completed — Lost to Follow-up | 2 | 2 | 1 | 1 | 0
Not completed — Covid quarantine | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TNM002 5 mg | TNM002 10 mg | TNM002 15 mg | HTIG | Placebo | Total
Number analyzed (Participants) | 61 | 61 | 29 | 59 | 30 | 240
Age, Continuous [Median (Full Range); unit: years of age] | 40 [20 to 62] | 38 [22 to 59] | 33 [22 to 62] | 36 [20 to 63] | 38.5 [19 to 60] | 38 [19 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 8 | 26 | 13 | 88
  Male | 41 | 40 | 21 | 33 | 17 | 152
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Anti-tetanus neutralizing antibody titers [Geometric Mean (Standard Deviation); unit: IU/mL] — Population: The administration of placebo precluded measurable antibody response generation, thus participants in the placebo group were excluded from the efficacy analyses regarding the changes in antibody titers. Baseline antibody titers were measured for placebo participants solely for demographic balance assessment and assay validation purposes.
  IU/mL | 0.4982 (2.1697) | 0.0916 (0.3253) | 0.0362 (0.0583) | 0.0596 (0.2530) | 0.0738 (0.2194) | 0.1782 (1.125)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Volunteers With an Increase of Anti-tetanus Neutralizing Antibody Titers Over Protective Level
Description: The increase of anti-tetanus neutralizing antibody titers were defined as ΔTiters, calculated as the post-administration antibody titers minus the baseline antibody titers. The antibody protective level is ΔTiters >0.01 IU/mL.
Time Frame: At 24 hours post-dose
Population: The analysis plan prespecified that placebo group data would not be collected for this outcome measure related to the anti-tetanus antibody level, as the administration of placebo precludes the generation of measurable antibody responses. Therefore, placebo recipients were analytically excluded from the efficacy analysis of antibody titer changes. The active control (HTIG) serves as the comparator for efficacy assessments, while the placebo group is retained solely for safety evaluations.
Measure: Count of Participants; unit: Participants
Arm/Group | TNM002 5 mg | TNM002 10 mg | TNM002 15 mg | HTIG | Placebo
Number analyzed (Participants) | 61 | 61 | 29 | 59 | 0
Participants | 56 | 61 | 29 | 48 | 0

2. Secondary Outcome: Change From Baseline in Anti-tetanus Neutralizing Antibody Titers (∆Titers)
Description: The increase of anti-tetanus neutralizing antibody titers were defined as ΔTiters, calculated as the post-administration antibody titers minus the baseline antibody titers. The antibody protective level is ΔTiters >0.01 IU/mL.
  The number of participants with evaluable anti-tetanus neutralizing antibody data were provided at each post-dose timepoint.
Time Frame: At 24 hours, 48 hours, and on Days 3, 7, 21, 30 and 90 post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | TNM002 5 mg | TNM002 10 mg | TNM002 15 mg | HTIG | Placebo
Number analyzed (Participants) | 61 | 61 | 29 | 59 | 0
IU/mL
  24 hours | 0.0450 [0.0338 to 0.0597] | 0.1095 [0.0844 to 0.1418] | 0.2094 [0.1637 to 0.2677] | 0.0200 [0.0158 to 0.0253] |
  48 hours | 0.0687 [0.0529 to 0.0889] | 0.1665 [0.1338 to 0.2071] | 0.3007 [0.2446 to 0.3695] | 0.0295 [0.0240 to 0.0362] |
  Day 3 | 0.0957 [0.0771 to 0.1188] | 0.2057 [0.1691 to 0.2503] | 0.3835 [0.3201 to 0.4593] | 0.0348 [0.0288 to 0.0419] |
  Day 7 | 0.1264 [0.1057 to 0.1511] | 0.2655 [0.2288 to 0.3081] | 0.4786 [0.4126 to 0.5551] | 0.0392 [0.0336 to 0.0456] |
  Day 21: number analyzed (Participants) | 60 | 61 | 29 | 59 | 0
  Day 21 | 0.1282 [0.1154 to 0.1425] | 0.2563 [0.2357 to 0.2788] | 0.3898 [0.3549 to 0.4280] | 0.0274 [0.0230 to 0.0327] |
  Day 30: number analyzed (Participants) | 59 | 60 | 29 | 58 | 0
  Day 30 | 0.1058 [0.0959 to 0.1166] | 0.2119 [0.1946 to 0.2306] | 0.3217 [0.2943 to 0.3518] | 0.0214 [0.0187 to 0.0243] |
  Day 90: number analyzed (Participants) | 58 | 60 | 28 | 58 | 0
  Day 90 | 0.0189 [0.0160 to 0.0223] | 0.0381 [0.0338 to 0.0430] | 0.0655 [0.0546 to 0.0785] | 0.0057 [0.0039 to 0.0080] |

3. Secondary Outcome: Proportion of Volunteers With an Increase of Anti-tetanus Neutralizing Antibody Titers Over Protective Level
Description: as for outcome 2
Time Frame: At 48 hours and on Days 3, 7, 21, 30, and 90 post-dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TNM002 5 mg | TNM002 10 mg | TNM002 15 mg | HTIG | Placebo
Number analyzed (Participants) | 61 | 61 | 29 | 59 | 0
Participants
  48 hours | 58 | 61 | 29 | 55 |
  Day 3 | 61 | 61 | 29 | 57 |
  Day 7 | 61 | 61 | 29 | 59 |
  Day 21: number analyzed (Participants) | 60 | 61 | 29 | 59 | 0
  Day 21 | 60 | 61 | 29 | 57 |
  Day 30: number analyzed (Participants) | 59 | 61 | 29 | 59 | 0
  Day 30 | 59 | 61 | 29 | 56 |
  Day 90: number analyzed (Participants) | 58 | 60 | 28 | 58 | 0
  Day 90 | 48 | 58 | 28 | 18 |

4. Secondary Outcome: Duration of Anti-tetanus Neutralizing Antibody Titers Increasing From Baseline Over Protective Level Post-dose
Description: as for outcome 2
Time Frame: Up to 105 (±7) days post dosing
Population: as for outcome 1
Measure: Median (Full Range); unit: Day
Arm/Group | TNM002 5 mg | TNM002 10 mg | TNM002 15 mg | HTIG | Placebo
Number analyzed (Participants) | 61 | 61 | 29 | 59 | 0
Day | NA [2 to 112] — More than half of the participants maintained antibody titers above protective level (0.01 IU/mL) through the end of the trial. | NA [58 to 111] — More than half of the participants maintained antibody titers above protective level (0.01 IU/mL) through the end of the trial. | NA [31 to 108] — More than half of the participants maintained antibody titers above protective level (0.01 IU/mL) through the end of the trial. | 59 [9 to 106] |

5. Secondary Outcome: Maximum Concentration (Cmax) of TNM002
Description: The peak serum concentration of TNM002 observed after administration.
Time Frame: Up to 105 days post dosing
Population: All TNM002-treated participants had evaluable post-dose concentration data for the calculation of Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | TNM002 5 mg | TNM002 10 mg | TNM002 15 mg
Number analyzed (Participants) | 61 | 61 | 29
ng/mL | 460 (57.6) | 967 (52.6) | 1710 (34.5)

6. Secondary Outcome: Time to Maximum Concentration (Tmax) of TNM002
Description: The time point at which the Cmax is observed following TNM002 administration.
Time Frame: Up to 105 days post dosing
Population: All TNM002-treated participants had evaluable post-dose concentration data for the calculation of Tmax.
Measure: Median (Full Range); unit: hours
Arm/Group | TNM002 5 mg | TNM002 10 mg | TNM002 15 mg
Number analyzed (Participants) | 61 | 61 | 29
hours | 312 [72 to 698] | 311 [72 to 698] | 144 [72 to 481]

7. Secondary Outcome: Elimination Half-life (t1/2) of TNM002
Description: The time required for the serum concentration of TNM002 to decrease by 50% during the elimination phase.
Time Frame: Up to 105 days post dosing
Population: Five participants were exlucded from the analysis due to model fitting failure for t1/2.
Measure: Median (Full Range); unit: hours
Arm/Group | TNM002 5 mg | TNM002 10 mg | TNM002 15 mg
Number analyzed (Participants) | 58 | 60 | 28
hours | 586 [415 to 988] | 596 [353 to 991] | 661 [416 to 867]

8. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to t (AUC0-t) of TNM002
Description: The total drug exposure of TNM002 over a defined time period (from administration to the last measurable concentration), calculated as the integral of the serum concentration-time curve.
Time Frame: Up to 105 days post dosing
Population: All TNM002-treated participants had evaluable post-dose concentration data for AUC analysis.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | TNM002 5 mg | TNM002 10 mg | TNM002 15 mg
Number analyzed (Participants) | 61 | 61 | 29
h*ng/mL | 524000 (231000) | 1080000 (384000) | 1810000 (499000)

9. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to ∞ (AUC0-∞) of TNM002
Description: The total systemic exposure of TNM002 from administration until complete elimination, calculated by combining AUC0-t and the extrapolated area from the last measurable concentration to infinity.
Time Frame: Up to 105 days post dosing
Population: Five participants were exlucded from the analysis due to model fitting failure for AUC0-∞.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | TNM002 5 mg | TNM002 10 mg | TNM002 15 mg
Number analyzed (Participants) | 58 | 60 | 28
h*ng/mL | 589000 (244000) | 1180000 (416000) | 1990000 (559000)

10. Secondary Outcome: Positive Rate of ADA in Volunteers in TNM002 Groups
Description: The proportion of participants who developed anti-drug antibodies (ADA) against TNM002 during the course of the trial.
Time Frame: Up to 105 days post dosing
Population: All TNM002-treated participants had evaluable post-dose immunogenicity data for the ADA analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | TNM002 5 mg | TNM002 10 mg | TNM002 15 mg
Number analyzed (Participants) | 61 | 61 | 29
Participants | 3 | 3 | 1

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 105 (±7) days post dosing
Description: The definition of adverse events in this trial is consistent with that specified in ClinicalTrials.gov.
  The causality assessment in this trial utilized a dichotomous classification: "Related" or "Not Related." For an adverse event of varying severity levels occurring in the same participant, the highest severity grade observed for that AE was used for analysis.
Arm/Group | TNM002 5 mg | TNM002 10 mg | TNM002 15 mg | HTIG | Placebo
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/61 | 0/29 | 0/59 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/61 | 0/29 | 1/59 | 0/30
Other Adverse Events (participants affected / at risk) | 30/61 | 29/61 | 14/29 | 32/59 | 16/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TNM002 5 mg (N=61) | TNM002 10 mg (N=61) | TNM002 15 mg (N=29) | HTIG (N=59) | Placebo (N=30)
Subdural hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TNM002 5 mg (N=61) | TNM002 10 mg (N=61) | TNM002 15 mg (N=29) | HTIG (N=59) | Placebo (N=30)
Blood triglycerides increased (Investigations) | 6 | 8 | 2 | 3 | 5
Blood uric acid increased (Investigations) | 6 | 7 | 0 | 4 | 2
Alanine aminotransferase (Investigations) | 2 | 1 | 2 | 2 | 4
Bilirubin conjugated increased (Investigations) | 1 | 4 | 0 | 4 | 0
Monocyte count increased (Investigations) | 1 | 2 | 1 | 3 | 0
Red blood cells urine positive (Investigations) | 3 | 0 | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 2 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 1 | 1 | 1
Blood cholesterol increased (Investigations) | 1 | 2 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 1 | 1 | 1
Blood glucose increased (Investigations) | 2 | 1 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 2 | 1 | 0 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 1 | 0 | 1 | 2
Lymphocyte count increased (Investigations) | 1 | 0 | 1 | 1 | 0
Thrombocyte count decreased (Investigations) | 1 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 2 | 0
Blood magnesium decreased (Investigations) | 0 | 1 | 0 | 2 | 2
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 0 | 1 | 2
Leukocytes urine positive (Investigations) | 0 | 0 | 1 | 1 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT05625477/Prot_SAP_000.pdf